CLINICAL TRIAL: NCT04263818
Title: Étude du Mouvement de l'opérateur et de l'Endoscope au Cours de la Coloscopie
Brief Title: Endoscopist and Endoscope Motions During Colonoscopy
Acronym: ScopeGuide
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IHU Strasbourg (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 19-003
Record Dates: First submitted 2020-02-07; First posted 2020-02-11 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Intestinal Disease; Colonic Diseases
Keywords: colonoscopy; tracking motion
MeSH Terms: conditions — Intestinal Diseases; Colonic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Motions during colonoscopy (Experimental): Recording of endoscopist and endoscope motions right after the endoscopic exam the patient came for
  Interventions: Procedure: Recording of endoscopist and endoscope motions right after the endoscopic exam the patient came for

INTERVENTIONS:
Procedure: Recording of endoscopist and endoscope motions right after the endoscopic exam the patient came for — Carrying out the endoscopic procedure planned for the patient with the dedicated colonoscope which has magnetic coils over the entire length of the insertion tube. These magnetic coils generate a pulsed magnetic field at low frequency. These pulses are transmitted to an external receiver, refreshed at 15 images per second, then relayed to the processor to generate a 3D representation of the colonoscope next to it of the endoscopic image. There is no additional risk to the patient compared to current practice.
  Recording of endoscopist and endoscope motions right after the endoscopic exam the patient came for.

SUMMARY:
The aim of the study is to record and analyze endoscopist and endoscope motions to identify key movements during colonoscopy.

DETAILED DESCRIPTION:
The increasing development of interventional digestive endoscopy raises the challenge to teach and learn complex endoscopic procedures. Nowadays experts are facing the challenge of explaining precisely an elaborate choreography of movements performed during the procedure, while novices are confronted with a broad range of hand, wrist and shoulder movements each resulting in different endoscope responses. The teaching strategy of endoscopy could benefit from a dedicated motion library that would associate the endoscopist's motion and the consequent endoscope response. A simplified endoscopic language made of individual motions could greatly shorten the learning curve.

The aim of the study is to record and analyze endoscopist and endoscope motions to identify key movements during colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patient male or female
* Patient over 18 years old
* Patient who are scheduled for a colonoscopy procedure under sedation
* Patient able to understand the study and provide written informed consent
* Patient affiliated to the French social security system.

Exclusion Criteria:

* Patient unable to provide a written informed consent
* Patient with an altered colonic anatomy due to previous surgery
* Patient with a known anomaly of the colon
* Patient carrying an implantable medical device (pacemaker…)
* Patient with a condition preventing its participation to study procedures, according to investigator's judgment
* Pregnancy or breastfeeding
* Patient in custody
* Patient under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-06-05 (Actual); Primary Completion 2021-06-05 (Actual); Study Completion 2021-07-05 (Actual)

PRIMARY OUTCOMES:
Body motions recording | At time of colonoscopy
  Body motions recording using the "Xsens" tracking device. The "Xsens" motion tracking system consists of 17 wireless motion sensors that are applied with straps to the endoscopist without hindering natural movements.
Endoscope motions recording | At time of colonoscopy
  Endoscope motions recording using the ScopeGuide tracking system. Real-time visualization of the ScopeGuide system is possible thanks to integrated electromagnetic coils and an external sensor that generate a 3D representation of the colonoscope next to the endoscopic image.
Endoscope wheels rotation recording | At time of colonoscopy
  External video recording of the endoscope wheels rotation
Endoluminal images recording | At time of colonoscopy
  Endoluminal images recording using the endoscopic camera.

CONTACTS AND LOCATIONS:
Overall Officials: Silvana PERRETTA, MD, PhD, Principal Investigator — Service de Chirurgie Digestive et Endocrinienne, NHC, Strasbourg
Locations (1):
- Service de Chirurgie Digestive et Endocrinienne, NHC, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaltenbach T, Leung C, Wu K, Yan K, Friedland S, Soetikno R. Use of the colonoscope training model with the colonoscope 3D imaging probe improved trainee colonoscopy performance: a pilot study. Dig Dis Sci. 2011 May;56(5):1496-502. doi: 10.1007/s10620-011-1614-1. Epub 2011 Mar 16. PMID 21409379